CLINICAL TRIAL: NCT03263754
Title: Do Patients With Chronic Obstructive Pulmonary Disease Engaging With Educational Films in Addition to Pulmonary Rehabilitation Gain Health-related Improvements?
Brief Title: Do Educational Digital Films Enhance Patient COPD Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aberystwyth University (Other)
Collaborators: Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10203918b3002e6f1be4a19987
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Pocket Medic; Behavioral: Pulmonary Rehabilitation
- Control (Active Comparator)
  Interventions: Behavioral: Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Pocket Medic — 10 short digital films utilising self-determination theory aiming to increase patient self-management
  Arms: Intervention
Behavioral: Pulmonary Rehabilitation — PR follows National Institute for Clinical Excellence guidelines delivering 14 sessions over 7 weeks utilising a multidisciplinary approach

SUMMARY:
This study aims to assess the efficacy of Pocket Medic to promote self-management and pulmonary rehabilitation adherence in COPD patients.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) refers to a group of lung conditions characterized by airways inflammation, small airways obstruction and progressive loss of lung function. There are 900,000 people diagnosed with COPD in England and Wales but allowing for under-diagnosis, the true prevalence could be 1.5 million. Sufferers are extensive health care users; where COPD is the second most common cause of emergency hospital admission in the United Kingdom with direct National Health Service costs over £800 million per year. Pulmonary Rehabilitation programs (PRPs) aim to provide education and support for patients whilst improving clinical outcomes, however, attendance to these programs can be low.

This study aims to trial a series of digital films aimed at educating patients about their condition from the comfort of their own home. Approximately 80 patients eligible for PR will be allocated to an experimental condition to receive a series of 10 digital films alongside their standard 7-week PR, solely to receive 10 digital films, or to a control condition in the form of standard PR (no digital films). Outcome measures such as PR attendance, hospital admissions, quality of life (QoL), disease knowledge, psychological need satisfaction and motivation will be measured pre and post. Analysis of this data between the experimental and control conditions pre-post intervention will provide useful information regarding the efficacy of digital film prescriptions as an adjunct to usual PR, or on its own, and the role this may play is encouraging PR attendance.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for pulmonary rehabilitation in Hywel Dda University Health Board.

Exclusion Criteria:

* Unwilling or unable to give informed consent
* life expectancy of less than 6 months
* unstable cardiovascular disease, dementia, cancers other than non-melanoma skins cancer
* any condition that precludes patients using laptops or mobile phones (e.g. blind, deaf)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Patient engagement | 10 weeks
  The level at which patients in the intervention arm watch the digital films
Patient Adherence | 10 weeks
  The level at which patients attend pulmonary rehabilitation sessions

SECONDARY OUTCOMES:
Disease Knowledge | 10 weeks and 6 months
  Scores on Bristol COPD Knowledge Questionnaire
Service Utilization | Baseline and 6 months
  Number of General Practioner visits and hospitalizations
Psychological self-management | 10 weeks and 6 months
  Patient scores on self-determination theory questionnaires modified to be relevant to COPD
Understanding COPD self-management | 10 weeks and 6 months
  Scores on the Understanding COPD self-management questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Liam Knox, Principal Investigator — Aberystwyth University
Locations (2):
- United Kingdom (2):
  - Glangwilli Hospital, Carmarthen, Carmarthenshire
  - Prince Phillip Hospital, Llanelli, Carmarthenshire

IPD SHARING:
Plan to Share IPD: No